CLINICAL TRIAL: NCT04612426
Title: the Effectiveness of Brain-computer Interface-pedaling Training System on Motor and Cognitive Function Rehabilitation of Stroke Patients
Brief Title: the Effectiveness of Brain-computer Interface-pedaling Training System on the Rehabilitation of Stroke
Acronym: BCI-PT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJUFH-R-001
Record Dates: First submitted 2020-10-28; First posted 2020-11-03 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2020-10

CONDITIONS: Rehabilitation; Stroke; Brain-computer Interface
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brain-computer Interface-Pedaling Training System (Experimental)
  Interventions: Device: Brain-computer Interface-Pedaling Training System
- Traditional Pedaling Training System (Sham Comparator): Patients wear the same EEG equipment that only collect data, but not guide training.
  Interventions: Device: Traditional Pedaling Training System

INTERVENTIONS:
Device: Brain-computer Interface-Pedaling Training System — The Brain-computer Interface-Pedaling Training System includes four parts: computer, monitor, EEG testing equipment and pedaling training equipment. The patient wears an EEG detection device, which calculates brain movement participation every 0.5 seconds. The system will provide real-time visual/auditory/somatosensory feedback to patients based on the results of participation, so that patients can participate in motor function training more attentively.
  Arms: Brain-computer Interface-Pedaling Training System
Device: Traditional Pedaling Training System — The patient will wear the same EEG equipment that will only collect data, but not guide training.
  Arms: Traditional Pedaling Training System

SUMMARY:
Stroke has become the first cause of death and disability among Chinese adults. 70%-80% of patients cannot live independently due to disability, which has brought a heavy burden to families, medical institutions and society. How to better evaluate and improve post-stroke motor and cognitive dysfunction has always been a hot research topic. With the rapid development of brain-computer interface technology, rehabilitation assessment based on quantitative EEG analysis is gradually being applied in the medical field. So we designed a brain-computer interface based on hierarchical task induction-pedaling rehabilitation training system to investigate the effectiveness on the rehabilitation of stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 40-80 years old；
* Patients with first ischemic stroke onset from 1 week to 3 months；
* Hemiplegia and cognitive impairment (Mini-Mental State Examination (MMSE) score <28 or Montreal Cognitive Assessment (MoCA) <25)；
* Consciousness, sitting balance level 1 or above, can cooperate with assessment and treatment;
* The patient or its authorized agent signs the informed consent form.

Exclusion Criteria:

* Severely impaired cognition, unable to pay attention to and understand screen information;
* Severe pain and limited mobility of lower extremity.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-02-10 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
The change of Fugl-Meyer motor function score of lower limbs | Two weeks after enrollment.
  The score range is 0-34 points, the higher the score, the better the motor function of lower limb.

SECONDARY OUTCOMES:
Attention index | Two weeks after enrollment.
  We used EEG equipment to calculate attention index which ranges 0-100 points. The higher the score, the higher the participation.
Digital Span Test (DST) | Two weeks after enrollment.
  The more correct numbers you recite, the greater your attention span.
Symbol Digit Modalities Test (SDMT) | Two weeks after enrollment.
  The more numbers converted, the better the ability to shift and maintain attention.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

REFERENCES:
- [Derived] Yuan Z, Peng Y, Wang L, Song S, Chen S, Yang L, Liu H, Wang H, Shi G, Han C, Cammon JA, Zhang Y, Qiao J, Wang G. Effect of BCI-Controlled Pedaling Training System With Multiple Modalities of Feedback on Motor and Cognitive Function Rehabilitation of Early Subacute Stroke Patients. IEEE Trans Neural Syst Rehabil Eng. 2021;29:2569-2577. doi: 10.1109/TNSRE.2021.3132944. Epub 2021 Dec 21. PMID 34871175